CLINICAL TRIAL: NCT01523262
Title: The Effect of Preconditioning to Prevent Perioperative Myocardial Ischemia in Elective Operation of Abdominal Aortic Aneurysm
Brief Title: Preventing Myocardial Ischemia by Preconditioning in Elective Operation for Abdominal Aortic Aneurysm
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Nikolaj Eldrup, MD, PHD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-20100012
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Aortic Aneurysm
Keywords: preconditioning; aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preconditioning and normal treatment (Active Comparator)
  Interventions: Procedure: preconditioning
- normal treatment (Placebo Comparator): Standard treatment
  Interventions: Procedure: Normal surgery, with sham intervention without inflating arm cuff

INTERVENTIONS:
Procedure: preconditioning — peripheral preconditioning induced by brief, intermittent constriction of blood supply to an arm
  Arms: Preconditioning and normal treatment
Procedure: Normal surgery, with sham intervention without inflating arm cuff
  Arms: normal treatment

SUMMARY:
Primary To investigate whether peripheral predonditioning induced by brief, intermittent constriction of blood supply to an arm can reduce the incidence of perioperative myocardial ischemia in patients operated electively for infrarenal aortic aneurysm.

Secondary To investigate the impact of peripheral preconditioning on perioperative inflammatory response.

To investigate whether peripheral preconditoning can protect against perioperative myocardial infarction and reduced cardiac pump function.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years, hospitalized for elective surgery of abdominal aortic aneurysm

Exclusion Criteria:

* Lack of informed consent.
* Hemiparetic patient.
* Pregnancy or nursing patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
measurements of CKMB and Troponin T | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aalborg Hospital, Aalborg, Aalborg
  - Aarhus University Hospital, Skejby, Aarhus, Aarhus N

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250